CLINICAL TRIAL: NCT03187717
Title: The Comparison of Total Intravenous Anesthesia and Inhalation Anesthesia Procedures Used in Oral and Maxillofacial Surgeries in View of Postoperative Complications and the Recovery Period
Brief Title: Total Intravenous Anesthesia and Inhalation Anesthesia
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ozlem Kocaturk, Medical doctor, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: OzlemKocaturk
Record Dates: First submitted 2017-05-22; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Complications
Keywords: Postoperative pain; Recovery period; Total intravenous anesthesia; Inhalation anesthesia
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIVA (Total intravenous anesthesia): Group TIVA; patients who used intravenous anesthesia procedure
- IA (Inhalation anesthesia): Group IA; patients who used inhalation anesthesia procedure

SUMMARY:
The aim of us is to define the incidence of postoperative complications and recovery time in view of two anesthesia procedures.

During the period between 01.01.2016 and 01.01.2017, totally 583 patients were included in the study, who had oral and maxillofacial surgeries. Anesthesia types were determined as total intravenous anesthesia (TIVA) and inhalation anesthesia (IA). Postoperative complications and recovery period were determined as tachycardia, bradycardia, hypertension, hypotension, recovery time, additional analgesia, nausea-vomiting. Both anesthesia procedures were compared in terms of these postoperative complications and recovery time.

DETAILED DESCRIPTION:
Totally American Society of Anesthesiologists (ASA) I-II, 18-60 ages, 583 patients who had had oral and maxillofacial operations for 30 minutes and over with TIVA and IA methods between 1st Jan, 2016 and 1st Jan, 2017. The ones who had insufficient data in their files and who were conscious / superficial sedation patients were excluded from the study. The patients were allocated to two groups as TIVA and IA. The total intravenous anesthesia group was named "Group TIVA" , and the volatile anesthesia group was named "Group IA".

All the patients were opened vascular access after being taken into the operation room and were given anesthesia induction with 1 µg/kg fentanyl, 2 mg/kg propofol and 0,8 mg/kg rocuronium. The patients in Group IA were given 1-2% volume sevoflurane in 50% oxygen and 50% nitrous oxide during maintenance of anesthesia, while the patients in group TIVA were applied 4-10 mg/kg/h propofol and 0.05-0.1 µg/kg fentanyl IV infusion with 50% oxygen and 50% air. While being woken up, each patient was given 0.3 mg/kg tenoxicam for analgesia and 0.2 mg/kg metoclopramide for nausea-vomiting prophylaxis in a routine way. Each patient was taken into recovery room after extubation and pulse rate, non-invasive blood pressure (NIBP) and oxygen saturation monitorization were done. Postoperative complication and vital finding tracks of each patient were done as usual and were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Totally American Society of Anesthesiologists (ASA) I-II, 18-60 ages patients who had had oral and maxillofacial operations for 30 minutes and over with TIVA and IA procedures between 1st Jan, 2016 and 1st Jan, 2017.

Exclusion Criteria:

* The ones who had insufficient data in their files and who were conscious/superficial sedation patients were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ASA I-II, 18-60 ages patients who had had maxillofacial surgery for 30 minutes and over with TIVA and IA prosedures between 1st Jan, 2016 and 1st Jan, 2017 were our study population.
Sampling Method: Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 1 year
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Kocaturk, MD, Principal Investigator — Faculty of Dentistry, Adnan Menderes University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gecaj-Gashi A, Hashimi M, Sada F, Baftiu N, Salihu S, Terziqi H, Bruqi B. Propofol vs isoflurane anesthesia-incidence of PONV in patients at maxillofacial surgery. Adv Med Sci. 2010;55(2):308-12. doi: 10.2478/v10039-010-0033-4. PMID 20934965
- [Background] Lee WK, Kim MS, Kang SW, Kim S, Lee JR. Type of anaesthesia and patient quality of recovery: a randomized trial comparing propofol-remifentanil total i.v. anaesthesia with desflurane anaesthesia. Br J Anaesth. 2015 Apr;114(4):663-8. doi: 10.1093/bja/aeu405. Epub 2014 Dec 10. PMID 25500679
- [Background] Jellish WS, Lien CA, Fontenot HJ, Hall R. The comparative effects of sevoflurane versus propofol in the induction and maintenance of anesthesia in adult patients. Anesth Analg. 1996 Mar;82(3):479-85. doi: 10.1097/00000539-199603000-00009. PMID 8623947
- [Background] Watson KR, Shah MV. Clinical comparison of 'single agent' anaesthesia with sevoflurane versus target controlled infusion of propofol. Br J Anaesth. 2000 Oct;85(4):541-6. doi: 10.1093/bja/85.4.541. PMID 11064611
- [Background] Bharti N, Chari P, Kumar P. Effect of sevoflurane versus propofol-based anesthesia on the hemodynamic response and recovery characteristics in patients undergoing microlaryngeal surgery. Saudi J Anaesth. 2012 Oct-Dec;6(4):380-4. doi: 10.4103/1658-354X.105876. PMID 23493938
- [Background] Adams HA, Schmitz CS, Baltes-Gotz B. [Endocrine stress reaction, hemodynamics and recovery in total intravenous and inhalation anesthesia. Propofol versus isoflurane]. Anaesthesist. 1994 Nov;43(11):730-7. doi: 10.1007/s001010050115. German. PMID 7840401
- [Background] Joo HS, Perks WJ. Sevoflurane versus propofol for anesthetic induction: a meta-analysis. Anesth Analg. 2000 Jul;91(1):213-9. doi: 10.1097/00000539-200007000-00040. PMID 10866915
- [Background] Dashfield AK, Birt DJ, Thurlow J, Kestin IG, Langton JA. Recovery characteristics using single-breath 8% sevoflurane or propofol for induction of anaesthesia in day-case arthroscopy patients. Anaesthesia. 1998 Nov;53(11):1062-6. doi: 10.1046/j.1365-2044.1998.00571.x. PMID 10023274